CLINICAL TRIAL: NCT00654563
Title: Memory Disorders Registry
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Dr. Robert Cohen, Ph.D., M.D., Cedars-Sinai Medical Center
Other Study IDs: IRB12126
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Dementia; Alzheimer's Disease; Parkinson Disease; Huntington Disease
Keywords: Memory Disorders; Memory loss; Age Associated Memory Impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Parkinson Disease; Huntington Disease; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The main Memory Disorders Registry only involves records-keeping to follow subjects' care, and does not involve any biospecimen collection. The optional postmortem exam (brain-only autopsy) obtains brain tissue, and it would be performed after death, so that no risks will impact the subject involved in the postmortem examination. With regard to cosmetic concerns, the incision is made from ear to ear through the neck region, leaving no disfiguration. The postmortem exam is not a genetic screen, but in rare instances it might find brain atrophy, although no specific inclusions. If found, the subject's family would be informed of this finding.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to collect data regarding the clinical course and outcome of patients suffering from memory disorders. Visits are charged to the individual's insurance inclusive of Medicare. Patients benefit from expert evaluation and treatment recommendations. Participants may be eligible for participation in experimental treatments in the future.

DETAILED DESCRIPTION:
The purpose of this long-term, observational patient outcome registry at Cedars-Sinai Medical Center is to collect information about subjects with memory disorders from their clinical care and treatment outcome(s). It plans to examine predictors of treatment outcomes among those individuals who enroll.

Currently, there are no curative treatments for memory disorders, and this study hopes to collect information on the disorders. Over the next 6 years, this registry expects to recruit 600 adults over the age of 18 who are concerned that they may have a memory problem, or who have been diagnosed with a memory problem such as occurs in Age Associated Memory Impairment, Alzheimer's disease, Vascular Dementia, Mixed Dementia, Dementia with Lewy Bodies, Frontotemporal Dementia, Parkinson's disease, or Huntington's disease.

The Memory Disorders Program owes its existence to patients agreeing to have their clinical information kept in a database for quality control and research purposes. This data will include physical and cognitive exams, laboratory tests and scans as well as information about their medications. Many potential subjects will call in with interest in our Memory Disorders Program, and a preliminary screening process will be performed over the phone. All potential subjects would be sent an informed consent document to look at before reviewing it with the study coordinator. Once they arrive at their initial visit, the research registry and its optional substudy (a postmortem exam available to all Cedars-Sinai patients) would be discussed with unlimited time for questions. If the subject, or his/ her surrogate decision maker (legally authorized representative, or LAR), consents to research, then his/ her clinical test results and (if applicable) the results of the postmortem exam will be kept on file for research purposes. If the subject/LAR consents, he/ she may also be contacted about any future research studies for which he/ she may be eligible. Patients who elect not to participate in this research will not be contacted for future studies. However, for those who are found to be ineligible and would like to learn about future studies as they arise, the Memory Disorders ICF offers them the option to be contacted in the future as new studies become available to them.

This research study will involve no collaborations, inside or outside of the Cedars-Sinai Medical Center. However, the subject's clinical care will involve collaborations with other departments within Cedars-Sinai Medical Center.

This registry will not involve any research-related costs, or any remunerative incentive.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Capable of providing informed consent and having a legal representative able to consent out of concern for future competency to consent (as defined by a Mini Mental State Exam score of <24) or capable of assent but incapable of giving competent informed consent, but with a legal representative able to provide informed consent
* Subject or family voices concern about their memory or possess knowledge that they have been diagnosed with a memory disorder such as Age Associated memory Impairment, Alzheimer's disease, Parkinson disease, Huntington disease, vascular dementia, mixed dementia, dementia with Lewy Bodies, or frontotemporal dementia

Exclusion Criteria:

* Children (less than 18 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Registry's study population will consist of private patients of Dr. Robert Cohen who have been diagnosed with a Memory Disorder or who are referred to him due to subjective reports of having a memory problem.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, Ph.D., M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States